CLINICAL TRIAL: NCT00002904
Title: PHASE I CLINICAL AND PHARMACOKINETIC STUDY TO DETERMINE THE SAFETY OF ECTEINASCIDIN-743 (ET-743) ADMINISTERED AS A SINGLE INTRAVENOUS INFUSION OVER 60 MINUTES EVERY 21 DAYS IN PATIENTS WITH SOLID TUMORS
Brief Title: Ecteinascidin 743 in Treating Adults With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-16951; EORTC-16951
Record Dates: First submitted 1999-11-01; First posted 2004-09-03 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Trabectedin

INTERVENTIONS:
Drug: trabectedin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of ecteinascidin 743 in treating adults with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the maximum tolerated dose (MTD) of ecteinascidin-743 (ET-743) when administered as a single intravenous infusion every 21 days in adults with solid tumors not amenable to standard therapy. II. Describe the qualitative and quantitative toxic effects of ET-743, and study the predictability, duration, intensity, onset, reversibility, and dose-relationship of these toxic effects in these patients. III. Propose a safe dose for a phase II study based on the MTD determined on this study. IV. Assess the pharmacokinetics of ET-743 at different dose levels. V. Document any antitumor effects of ET-743 in these patients.

OUTLINE: This is a multicenter study. All patients receive ET-743 IV over 3 hours every 21 days for 4 courses. Treatment continues in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of ET-743 until the maximum tolerated dose is determined. Patients are followed at 1 month, then every 3 months until disease progression.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study over 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed solid tumor that is not amenable to standard therapy No evidence of brain involvement or leptomeningeal disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: ANC at least 2,000/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL Hepatic: Bilirubin less than 1.5 mg/dL Transaminases normal (no greater than 2.5 times normal if liver metastases) Alkaline phosphatase normal (no greater than 2.5 times normal if liver or bone metastases) No history of chronic liver disease, e.g., chronic active hepatitis, cirrhosis Renal: Creatinine no greater than 1.4 mg/dL Creatinine clearance at least 60 mL/min Other: No active bacterial infection (e.g., abscess) or with fistulae No grade 2 or worse neurotoxicity No concurrent medical condition that precludes treatment No history of alcoholism, drug addiction, or psychotic disorder Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Colony-stimulating factors allowed for specific indications At least 4 weeks since prior biologic therapy, immunotherapy, or growth factors Chemotherapy: No prior intensive chemotherapy with bone marrow or stem cell support At least 4 weeks since chemotherapy (6 weeks since nitrosoureas, mitomycin, or high-dose carboplatin) Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since radiotherapy Concomitant palliative local radiotherapy allowed for existing lesion Surgery: Recovered from prior surgery Other: No concurrent investigational drug Concurrent prophylactic antiemetics allowed after first therapy course

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1996-02

CONTACTS AND LOCATIONS:
Overall Officials: Chris Twelves, MD, BMedSci, FRCP, Study Chair — University of Glasgow
Locations (49):
- Ludwig Boltzmann - Institute for Applied Cancer Research, Vienna (Wien), Austria
- Belgium (3):
  - Institut Jules Bordet, Brussels (Bruxelles)
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Herlev Hospital - University Hospital of Copenhagen, Herlev
- France (14):
  - Institut Bergonie, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges-Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - CHU de la Timone, Marseille
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Institut Curie - Section Medicale, Paris
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut Claudius Regaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Hopital Paul Brousse, Villejuif
  - Institut Gustave Roussy, Villejuif
- Germany (4):
  - Martin Luther Universitaet, Halle
  - Universitats-Krankenhaus Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum Nurnberg, Nuremberg (Nurnberg)
- University of Ioannina, Ioannina, Greece
- Israel (2):
  - Rambam Medical Center, Haifa
  - Schneider Children's Medical Center of Israel, Petah Tikva
- Italy (5):
  - Centro di Riferimento Oncologico - Aviano, Aviano
  - Istituto Europeo Di Oncologia, Milan
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Naples (Napoli)
  - San Raffaele Hospital, Rome
  - Istituti Fisioterapici Ospitalieri - Roma, Rome
- Netherlands (5):
  - Academisch Ziekenhuis der Vrije Universiteit, Amsterdam
  - Antoni van Leeuwenhoekhuis, Amsterdam
  - Academisch Ziekenhuis Groningen, Groningen
  - St. Radboud University Hospital, Nijmegen
  - Rotterdam Cancer Institute, Rotterdam
- Norwegian Radium Hospital, Oslo, Norway
- Instituto Portugues de Oncologia de Francisco Gentil, Lisbon, Portugal
- Hospital Universitario 12 de Octubre, Madrid, Spain
- Switzerland (5):
  - University Hospital, Basel
  - Ospedale San Giovanni, Bellinzona
  - Inselspital, Bern, Bern
  - Clinique De Genolier, Genolier
  - Kantonsspital - Saint Gallen, Sankt Gallen
- United Kingdom (4):
  - Royal Marsden NHS Trust, London, England
  - Newcastle General Hospital, Newcastle upon Tyne, England
  - Western General Hospital, Edinburgh, Scotland
  - Beatson Oncology Centre, Glasgow, Scotland